CLINICAL TRIAL: NCT04558684
Title: Short Course Radiotherapy With Total Neoadjuvant Chemotherapy and Immunotherapy in Rectal Cancer
Brief Title: Radiotherapy With Neoadjuvant Chemotherapy and Immunotherapy in Rectal Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inadequate patient enrollment
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Chief of gastrointestinal oncology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WUGO-002
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Rectal Cancer; Radiotherapy; Immunotherapy; Organ Preservation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy, chemotherapy and PD1 inhibitor (Experimental): Treatment will comprise 5 daily fractions of radiotherapy at 5 Gy per fraction followed by chemotherapy and immunotherapy. Those who achieve a clinical complete response will be considered for organ preservation approach. All other patients will receive standard surgery.
  Interventions: Drug: Chemotherapy; Drug: Immunotherapy; Radiation: IMRT

INTERVENTIONS:
Drug: Chemotherapy — CAPOX (6 cycles): Oxaliplatin(130mg/m2) on day 1 of each cylce and Capecitabine: Dose of 2000mg/m2,14 days, q3w
Drug: Immunotherapy — Camrelizumab (6 cycles): 200mg on day 1 of each cycle, q3w
Radiation: IMRT — Radiotherapy (5 Gy x 5 fractions)

SUMMARY:
This is a open-label, single-arm study to investigate the safety and efficacy of Total neoadjuvant chemotherapy with camrelizumab, an anti-PD-1 antibody drug following short course radiotherapy in patients with rectal cancer.

DETAILED DESCRIPTION:
Patients with rectal cancer are assigned to receive preoperative 5 × 5 Gy irradiation over 5 days with total neoadjuvant chemotherapy and camrelizumab, an anti-PD-1 antibody drug. The Primary Objective is to assess clinical complete response of an organ preservation approach and the secondary objective to assess safety in all enrolled patients, local regrowth rate and other cancer specific outcomes (metastasis-free survival, colostomy-free survival and overall survival), longitudinal health-related quality of life of this organ preservation approach.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who personally provided written consent for participation in the study
2. Treatment-naive patients with rectal cancer, in whom the inferior margin of the tumor is at a distance of 10 cm or less from the AV before CRT
3. Histologically confirmed adenocarcinoma of rectum (non-metastatic, >T2N0 or low T2N0 rectal cancer) not eligible for up-front organ preservation surgery as deemed by multidisciplinary evaluation
4. Patients with the ECOG performance status of 0 or 1 at the time of enrollment
5. Women of childbearing potential who consent to practicing contraception during the period from giving informed consent to at least 23 weeks after the last dose of therapy
6. Male patients who consent to practicing contraception during the period from giving informed consent to at least 31 weeks after the last dose of the study drug
7. Patients must have acceptable organ and marrow function as defined below:

Absolute neutrophil count (ANC) >1,500/uL Hg > 8.0 g/dL; if blood transfusion is performed for achieving adequate hemoglobin level, the level should stay above goal for at least 1 week after transfusion Platelets >100,000/uL Total bilirubin <1.5X normal institutional limits aspartate aminotransferase (AST) (SGOT) / alanine aminotransferase (ALT)(SGPT) < 3X upper limit of normal Creatinine <1.5X upper limit of normal or creatinine clearance (CrCL)>50 by Cockcroft-Gault

Exclusion Criteria:

1. Patients with recurrent rectal cancer or a history of pelvic radiation
2. Patients with a history of inflammatory bowel disease
3. Patients with a history of pneumonitis or interstitial lung disease
4. Patients with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease
5. Patients requiring treatment with systemic corticosteroids or immunosuppressants or who have received these treatments within 14 days before enrollment in the study
6. Patients with a history of thyroid dysfunction
7. Patients with a history or finding of cardiovascular risk
8. Patients who are positive for any of the following: HIV1 antibody, HIV2 antibody, HTLV1 antibody
9. Patients who are pregnant or lactating or who may be pregnant
10. Patients with significant unstable mental diseases or other medical diseases that may interfere with the safety of the subjects, obtaining informed consent, or compliance with the procedures for the clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response rate (cCR) | 8 (+/-4 ) weeks
  Proportion of patients who achieve a clinical complete response following treatment

SECONDARY OUTCOMES:
Local regrowth rate | 2 year
  Presence of adenocarcinoma within the rectal wall or within the mesorectum confirmed by pathology
Disease free survival (DFS) | 5 year
  Five years disease-free survival of this group of patients
Overall survival (OS) | 5 year
  Fives years overall survival of this group of patients
Incidence of adverse events (AEs) | 1 year
  Incidence of adverse events will be assessed according to the latest "Clavien- Dindo Classification of surgical complications" and Common Terminology Criteria of Adverse Events (CTCAE).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China